CLINICAL TRIAL: NCT03014141
Title: The Effect of Oat Bran on Bowel Function and Appetite. A Randomized, Double-blind, Placebo-controlled, Cross-over Intervention Study in Healthy Humans.
Brief Title: Effect of Oat Bran on Bowel Function and Appetite
Acronym: OATGUT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study supply issues
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2015-12-10-OAT
Record Dates: First submitted 2016-12-21; First posted 2017-01-09 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Gastrointestinal Disorder, Functional
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oat bran (Oatwell 28) (Active Comparator): A beverage containing 11 gram (3 gram of oat beta-glucan) of Oat bran (Oatwell 28) will be consumed before breakfast
  Interventions: Other: Oat bran (Oatwell 28)
- Maltodextrin (Placebo Comparator): A beverage containing 11 gram of maltodextrin will be consumed before breakfast.
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Other: Oat bran (Oatwell 28) — 11 g oat bran containing 3.1 gram oat beta-glucan
  Other Names: Oat bran oat beta-glucan
  Arms: Oat bran (Oatwell 28)
Other: Maltodextrin — 11 g of Maltodextrin
  Arms: Maltodextrin

SUMMARY:
The consumption of oat bran fiber also has a significant bulking effect in humans. However, besides fecal bulk, dietary fiber can promote gut health in other ways. Therefore, the purpose of this study is to investigate the effects of oat bran (rich in oat beta-glucan) supplementation on bowel function and appetite.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo-controlled crossover study it involves a total of 8 visits with a 14 day run-in period for total study duration of 84 days. A washout period of 2 weeks will occur in between the 2, 28 day treatment periods. The effects of an oat bran beverage for breakfast on bowel function will be tested after 2 week and 4 weeks of intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female between the ages of 18-60 years
* Subject has a body mass index of ≥18.5 and ≤30 kg/m2 at screening visit.
* Subject is willing to stick to their normal habitual diet excluding the consumption of any unusual high energy-rich or fat-rich meals or prolonged fasting, etc. through the study period.
* Subject is willing to maintain their habitual physical activity patterns throughout the study period.
* Subject has been weight stable within the last 6 months.
* Subject has no health conditions that would prevent him or her from fulfilling the study requirements as judged by the investigator on the basis of medical history and routine laboratory test results.
* Low fiber consumer (≤14 g per day)
* Subject is willing to follow study procedures and dietary restrictions (ex: stick to habitual diet, refrain from consuming alcohol 24 hours prior to test days).

Exclusion Criteria:

* History of a gastrointestinal disorder
* Lactose intolerant
* High fiber consumer (≥15 g per day)
* Use of pre-and probiotics in the past 90 days
* High protein consumer (i.e. vegetarians or those who follow diets high in protein such as paleo)
* History of psychological illness or conditions that may interfere with subjects ability to understand study directions
* Use of antibiotics or signs of active systemic infection in the last 6 months.
* Subjects who are on hypo/hypercaloric diet aiming for weight loss or weight gain
* History or presence of cancer in the prior 2 years (except for non-melanoma skin cancer).
* Currently pregnant, lactating or planning to be pregnant during the study period
* Regular use of dietary supplements (ex: fish oil, riboflavin, etc.), 90 days prior to study inclusion
* Exposure to any non-registered drug product within the last 30 days prior to screening visit
* History of or strong potential for alcohol or substance abuse (within 12 months of screening visit). Alcohol abuse is defined as >60g (men)/40g (women) pure alcohol per day (1.5 L/ 1 l beer resp. 0.75l/0.5l wine).
* Allergy or sensitivity to oat bran or any meals or snacks provided
* Current smoker or use of tobacco products in the past 90 days
* Concurrent or recent participation (30 days) in a dietary intervention trial
* Anything in the judgment of the investigator would interfere with the subject's ability to comply with the study (protocol), which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Whole gut transit time | 4 weeks
  Whole gut transit time is the time required for the passage of 80% of radio-opaque markers (ROM) which are detected by x-ray in the fecal samples collected over the next 5 days after swallowing the ROM.

SECONDARY OUTCOMES:
Whole gut transit time | 2 weeks
  Whole gut transit time is the time required for the passage of 80% of radio-opaque markers (ROM) which are detected by x-ray in the fecal samples collected over the next 5 days after swallowing the ROM.
Stool frequency | 2 weeks and 4 weeks
  using a bowel movement diary
Fecal output | 2 weeks and 4 weeks
  Fecal out is the weight of the fecal samples collected over the 5 days preceding the 2 week and 4 week time point
Percent fecal moisture | 2 weeks and 4 weeks
  Fecal moisture is determined by freeze drying fecal samples and calculating the percent moisture in the fecal sample
Bristol Stool Score | 2 weeks and 4 weeks
  using Bristol Stool Chart
Fecal pH | 2 weeks and 4 weeks
Subjective measures of bowel comfort | 2 weeks and 4 weeks
  Gastrointestinal Quality of life questionnaires (GIQLI)
Gut microbiota | 2 weeks and 4 weeks
  Using 16S ribosomal RNA sequencing techniques
Fecal short chain fatty acids | 2 weeks and 4 weeks
  Using gas chromatography
Fecal total bile acids | 2 weeks and 4 weeks
Fecal enzymes | 2 weeks and 4 weeks
  fecal beta-glucoronidase
Fecal ammonia | 2 weeks and 4 weeks
Intestinal gas production | 2 weeks and 4 weeks
  using breath hydrogen production
Appetite | 2 weeks and 4 weeks
  Appetite will be measured via visual analogue score (VAS)
Ad libitum energy intake | 2 weeks and 4 weeks
  Ad libitum energy intake is measured by serving the subject an excess of food

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Slavin, PhD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grabitske HA, Slavin JL. Low-digestible carbohydrates in practice. J Am Diet Assoc. 2008 Oct;108(10):1677-81. doi: 10.1016/j.jada.2008.07.010. PMID 18926133
- [Background] Stewart ML, Nikhanj SD, Timm DA, Thomas W, Slavin JL. Evaluation of the effect of four fibers on laxation, gastrointestinal tolerance and serum markers in healthy humans. Ann Nutr Metab. 2010;56(2):91-8. doi: 10.1159/000275962. Epub 2010 Jan 19. PMID 20090313
- [Background] Chen HL, Haack VS, Janecky CW, Vollendorf NW, Marlett JA. Mechanisms by which wheat bran and oat bran increase stool weight in humans. Am J Clin Nutr. 1998 Sep;68(3):711-9. doi: 10.1093/ajcn/68.3.711. PMID 9734752